CLINICAL TRIAL: NCT00198679
Title: Effect of Chlorhexidine Skin Cleansing on Skin Flora of Newborn Infants in Bangladesh
Brief Title: Effect of Chlorhexidine Skin Cleansing on Skin Flora
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H.22.03.10.07.A2
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2006-05

CONDITIONS: Skin Diseases, Infectious
Keywords: skin cleansing; Bangladesh; Skin Flora; Newborn; infectious disease; chlorhexidine
MeSH Terms: conditions — Skin Diseases, Infectious; Communicable Diseases | interventions — Chlorhexidine

INTERVENTIONS:
Drug: Chlorhexidine

SUMMARY:
Given the potential of skin cleansing with chlorhexidine as a safe, feasible, and cost-effective intervention for reducing neonatal death in developing country settings, this study follows a trial already underway in Nepal to test the impact of a single cleansing of the skin with baby wipes cotaining chlorahexidine.

DETAILED DESCRIPTION:
This study is designed to test the impact of a single cleansing of the skin with 0.25% or 4.0% Chlorhexidine wipes on qualitative and quantitative skin flora and skin condition in newborn infants. The study takes place in the Special Care Nursery at Dhaka Shishu Hospital in Dhaka, Bangladesh.

ELIGIBILITY:
Inclusion Criteria:

* Infant admitted to Special Care Nursery at Dhaka Shishu Hospital less than 48 hours chronological age
* parental consent must be obtained

Exclusion Criteria:

* infants being admitted for major surgical procedure which is attended by high rate of infectious complications
* sepsis
* clinically-evident skin infection
* generalized skin disease
* structural defect of the skin involving greater than 5% of the body surface
* with a major congenital anomaly
* with a known immunodeficiency

Max Age: 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210
Dates: Start 2004-03; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Wiping of newborn skin will be done immediatly upon enrollment in study, with follow up during hosptial stay and up to two weeks to determine skin condition and presence of any kind of skin infection.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Darmstadt, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Dhaka Shishu Hospital, Dhaka, Bangladesh